CLINICAL TRIAL: NCT06971640
Title: Advancing Identification of Circadian Delay in ADHD Youth: Associations With Clinical Heterogeneity and Cognition
Acronym: CIRCA
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00116918; R01MH136425 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-05-14 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-05

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity; ADHD
Keywords: ADHD; attention deficit disorder with hyperactivity; circadian rhythm; dim light melatonin onset
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Salivary melatonin will be collected. Eleven ~2ml saliva samples will be collected, one every 30 minutes, over a 5 hour period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to better understand sleep and circadian functioning in children with ADHD using home-based measures, parent report, and a lab based melatonin assessment. Investigators will also examine how sleep relates to psychiatric health and cognition among children with ADHD. The investigator for this study is Dr. Jessica Lunsford-Avery from the Department of Psychiatry.

DETAILED DESCRIPTION:
Participants will be asked to review and sign a consent form to enroll. As part of the study, participants will:

* Attend three study visits where they will be asked to complete questionnaires and assessments related to their child's attention and behavior, psychiatric health, and sleep habits. One of these visits is a lab-based melatonin assessment at night.
* Be asked to have their child wear a device (similar to a wrist watch) for a 7-day period. Parents will also be asked to complete an electronic daily diary about their child's sleep.
* Be asked to have their child wear a skin temperature sensor each evening after dinner until they wake up the next morning.
* Be asked to use a mattress sensor which measures movement, sleep state, and heart rate.

Participants will be compensated for their time.

ELIGIBILITY:
Inclusion Criteria:

1. Child ages 6-9
2. Meet criteria for a primary psychiatric diagnosis of DSM-5 ADHD, any presentation
3. Intellectual functioning >80
4. Healthy (i.e., no major medical problems)
5. If applicable, willingness to suspend use of melatonin during the study period

Exclusion Criteria:

1. Meet DSM-5 criteria for psychosis, bipolar, or autism spectrum disorders
2. Diagnosis of occult sleep disorders, including sleep apnea or restless leg syndrome
3. Medication for sleep other than melatonin
4. Plans to initiate stimulant medication during the study period

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with ADHD ages 6-9 in the Duke University Health System
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Circadian Rhythm (Sleep Timing) | Nightly for 7 nights (at-home assessment)
  Wearable sensor data collection includes 3 sensors and supporting materials. The GreenTEG Core sensor will measure changes in core body temperature (CBT) beginning each evening and continuing through the night until morning waking. The Withings Mat will index times in/out of bed and related sleep metrics. The Garmin Vivosmart 5 will continuously measure movement and heart rate.
DLMO - Dim Light Melatonin Onset | Day 8 (second in-person study visit)
  Salivary melatonin will be collected during an in-lab assessment, occurring on Friday night following the home assessment. Eleven saliva samples (~2ml) will be collected in a darkened environment every 30 min for a period beginning 4 hours before the child's average weeknight bedtime and extending to 1 hour after their average weeknight bedtime as verified by the previous week's sleep diary. The time at which salivary melatonin concentrations exceed 4 pg/mL will be used for determining DLMO. Circadian alignment will be measured via phase angle calculation, or the duration of time between DLMO and average bedtime as recorded by (1) sleep diary and (2) average sleep onset (actigraphy).

SECONDARY OUTCOMES:
Sleep disturbances as measured by parent report Children's Sleep Habits Questionnaire (CSHQ) | Immediately following the study period (up to approximately 2 weeks)
  Total score is the sum of all the scored questions on the CSHQ. The score ranges from 33 to 99, where a score above 41 indicates a pediatric sleep disorder.
Sleep routines as measured by the Pediatric Sleep Practices Questionnaire (PSPQ) | Immediately following the study period (up to approximately 2 weeks)
  The PSPQ provides information about sleep timing and consistency of sleep timing across weekends versus weekdays. The total score is standardized to a T-score with a mean of 50 and a standard deviation of 10.
Chronotype will be measured by parent report Children's Chronotype Questionnaire (CCTQ) | Immediately following the study period (up to approximately 2 weeks)
  Chronotypes are natural preferences of the body for wakefulness and sleep. Morning to Evening (M/E) scale-scores range from 10 (extreme morningness) to 49 (extreme eveningness). Morning types are classified by a M/E scale score of ≤23, intermediate types by a score of 24-32, and evening types by a score ≥33.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Lunsford-Avery, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
RTI International will be involved in deidentified data analysis.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be accessible by researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals and questions for data access should be directed to NDAHelp@mail.nih.gov. To gain access, data requestors will need to sign a data access agreement at https://nda.nih.gov/nda/access-data-info.html.
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Yektas C, Tufan AE, Sarigedik E. Sleep habits of children diagnosed with attention/ deficit/ hyperactivity disorder and effects of treatment on sleep related parameters. Asian J Psychiatr. 2020 Aug;52:102045. doi: 10.1016/j.ajp.2020.102045. Epub 2020 Apr 9. PMID 32361211
- [Background] Becker SP, Langberg JM, Eadeh HM, Isaacson PA, Bourchtein E. Sleep and daytime sleepiness in adolescents with and without ADHD: differences across ratings, daily diary, and actigraphy. J Child Psychol Psychiatry. 2019 Sep;60(9):1021-1031. doi: 10.1111/jcpp.13061. Epub 2019 Apr 29. PMID 31032953
- [Background] Merikanto I, Lahti J, Kuula L, Heinonen K, Raikkonen K, Andersson S, Strandberg T, Pesonen AK. Circadian preference and sleep timing from childhood to adolescence in relation to genetic variants from a genome-wide association study. Sleep Med. 2018 Oct;50:36-41. doi: 10.1016/j.sleep.2018.04.015. Epub 2018 Jun 1. PMID 29982088
- [Background] Dalsgaard S, Ostergaard SD, Leckman JF, Mortensen PB, Pedersen MG. Mortality in children, adolescents, and adults with attention deficit hyperactivity disorder: a nationwide cohort study. Lancet. 2015 May 30;385(9983):2190-6. doi: 10.1016/S0140-6736(14)61684-6. Epub 2015 Feb 26. PMID 25726514
- [Background] Peasgood T, Bhardwaj A, Biggs K, Brazier JE, Coghill D, Cooper CL, Daley D, De Silva C, Harpin V, Hodgkins P, Nadkarni A, Setyawan J, Sonuga-Barke EJ. The impact of ADHD on the health and well-being of ADHD children and their siblings. Eur Child Adolesc Psychiatry. 2016 Nov;25(11):1217-1231. doi: 10.1007/s00787-016-0841-6. Epub 2016 Apr 1. PMID 27037707
- [Background] Chhibber A, Watanabe AH, Chaisai C, Veettil SK, Chaiyakunapruk N. Global Economic Burden of Attention-Deficit/Hyperactivity Disorder: A Systematic Review. Pharmacoeconomics. 2021 Apr;39(4):399-420. doi: 10.1007/s40273-020-00998-0. Epub 2021 Feb 8. PMID 33554324
- [Background] Libutzki B, Ludwig S, May M, Jacobsen RH, Reif A, Hartman CA. Direct medical costs of ADHD and its comorbid conditions on basis of a claims data analysis. Eur Psychiatry. 2019 May;58:38-44. doi: 10.1016/j.eurpsy.2019.01.019. Epub 2019 Feb 22. PMID 30802682
- [Background] Doshi JA, Hodgkins P, Kahle J, Sikirica V, Cangelosi MJ, Setyawan J, Erder MH, Neumann PJ. Economic impact of childhood and adult attention-deficit/hyperactivity disorder in the United States. J Am Acad Child Adolesc Psychiatry. 2012 Oct;51(10):990-1002.e2. doi: 10.1016/j.jaac.2012.07.008. Epub 2012 Sep 5. PMID 23021476
- [Background] Sibley MH, Arnold LE, Swanson JM, Hechtman LT, Kennedy TM, Owens E, Molina BSG, Jensen PS, Hinshaw SP, Roy A, Chronis-Tuscano A, Newcorn JH, Rohde LA; MTA Cooperative Group. Variable Patterns of Remission From ADHD in the Multimodal Treatment Study of ADHD. Am J Psychiatry. 2022 Feb;179(2):142-151. doi: 10.1176/appi.ajp.2021.21010032. Epub 2021 Aug 13. PMID 34384227
- [Background] Zhao X, Page TF, Altszuler AR, Pelham WE 3rd, Kipp H, Gnagy EM, Coxe S, Schatz NK, Merrill BM, Macphee FL, Pelham WE Jr. Family Burden of Raising a Child with ADHD. J Abnorm Child Psychol. 2019 Aug;47(8):1327-1338. doi: 10.1007/s10802-019-00518-5. PMID 30796648
- [Background] Xu G, Strathearn L, Liu B, Yang B, Bao W. Twenty-Year Trends in Diagnosed Attention-Deficit/Hyperactivity Disorder Among US Children and Adolescents, 1997-2016. JAMA Netw Open. 2018 Aug 3;1(4):e181471. doi: 10.1001/jamanetworkopen.2018.1471. PMID 30646132